CLINICAL TRIAL: NCT01446250
Title: A Randomized, Open Label Trial of the Safety and Efficacy of DEB025/Alisporivir in Combination With Pegylated Interferon-α2a and Ribavirin (Peg-INFα2a/RBV) and Boceprevir in Combination With Peg-INFα2a/RBV in African American Treatment-naïve Patients With Chronic Hepatitis C Genotype 1
Brief Title: Alisporivir (Deb025) and Boceprevir Triple Therapies in African American Participants Not Previously Treated for Chronic Hepatitis C Genotype 1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDEB025A2307
Record Dates: First submitted 2011-09-26; First posted 2011-10-05 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C
Keywords: Chronic hepatitis C; Cyclophilin inhibitor
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — alisporivir; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2a; Ribavirin

ARMS (2):
- Alisporivir (Experimental): At the time of partial clinical hold, participants randomized to original treatment arms A and B (Alisporivir triple therapy arms with Peginterferon alfa-2a and Ribavirin) discontinued alisporivir treatment immediately while continuing their treatments with the other two therapies. These participants were combined into the same arm because they received the same dose of alisporivir 400 mg twice per day (BID) for the same duration. Amendment 1 offered them the opportunity to continue in the study receiving boceprevir triple therapy.
  Interventions: Drug: Alisporivir; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Boceprevir (Active Comparator): Participants randomized to boceprevir triple therapy with Peginterferon alfa-2a and Ribavirin (the original treatment arm C).
  Interventions: Drug: Boceprevir; Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Alisporivir — ALV 200 mg soft gel capsules administered orally
  Other Names: DEB025
  Arms: Alisporivir
Drug: Boceprevir — BOC 800 mg (4 x 200 mg soft gel capsules) administered orally
  Other Names: Victrelis®
  Arms: Boceprevir
Drug: Peginterferon alfa-2a — PEG 180 μg administered via subcutaneous (s.c.) injection once weekly
  Other Names: Pegasys®
Drug: Ribavirin — RBV 200 mg tablets (weight-based dose: < 75 mg = 1000 mg/day; ≥ 75 kg = 1200 mg/day) administered orally in a divided daily dose
  Other Names: Copegus®

SUMMARY:
This study will assess the safety and efficacy of alisporivir (ALV) and boceprevir (BOC), each in combination with Peginterferon alfa-2a (PEG) and Ribavirin (RBV), in African American participants who have never received treatment for their chronic hepatitis C (HCV) genotype 1 infection.

ELIGIBILITY:
Inclusion criteria:

* Chronic HCV genotype 1 infection
* No previous treatment for HCV infection
* African American ethnicity
* Serum HCV RNA ≥ 1000 IU/ml, assessed by quantitative polymerase chain reaction or equivalent at screening visit, no upper limit
* A liver biopsy within 3 years prior to baseline

Exclusion criteria:

* HCV genotype different from genotype 1 or co-infection with other HCV genotype
* Co-infection with Hepatitis B or HIV
* Any other cause of relevant liver disease other than HCV
* Presence or history of hepatic decompensation
* Alanine aminotransferase (ALT) ≥ 10 times ULN, more than 1 episode of elevated bilirubin (> ULN) in past 6 months

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigational Site, Beverly Hills, California
  - Novartis Investigational Site, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Alisporivir: Participants randomized to Treatment A and B received Alisporivir (ALV) 400 mg twice daily (BID) with Peginterferon alfa-2a (PEGinf) and Ribavirin (RBV) in Treatment Period 1.
- Boceprevir: Participants randomized to Treatment C received Boceprevir (BOC) 800 mg three times daily (TID) with PEGinf and RBV in Treatment Period 1. Participants who received ALV in Treatment Period 1 and were put on clinical hold for 4 weeks, received BOC 800 mg TID with PEGinf and RBV in Treatment Period 2.
- PEGinf + RBV: Participants who received ALV in Treatment Period 1 were put on clinical hold but continued receiving PEGinf and RBV for 4 weeks, after which they switched to BOC triple therapy in Treatment Period 2.
- No Intervention: Participants who had an End of Treatment Response (ETR) were followed-up for 24 weeks after the last dose of BOC triple therapy (in Treatment Period 2) and participants who did not respond for any reason or discontinued the treatment early were followed-up for 12 weeks after the last dose of BOC (in Treatment Period 2).
Period: Treatment Period 1
Arm/Group | Alisporivir | Boceprevir | PEGinf + RBV | No Intervention
Started | 5 | 3 | 0 | 0
Completed | 5 | 2 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Period: Clinical Hold
Arm/Group | Alisporivir | Boceprevir | PEGinf + RBV | No Intervention
Started | 0 | 2 | 5 | 0
Completed | 0 | 2 | 5 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Alisporivir | Boceprevir | PEGinf + RBV | No Intervention
Started | 0 | 7 | 0 | 0
Completed | 0 | 6 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Period: Follow-up
Arm/Group | Alisporivir | Boceprevir | PEGinf + RBV | No Intervention
Started | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- All Enrolled Participants: Analysis was performed on all enrolled participants.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Discontinued Study Drug or Required Dose Reduction or Dose Interruption Due to Treatment-emergent Adverse Events
Time Frame: within 48 weeks
Population: No data has been reported because planned data analyses were not performed as the study was terminated before the outcome measure time point.
Arm/Group | Alisporivir | Boceprevir
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Emergence of Resistant Mutations
Time Frame: within 48 weeks
Population: as for outcome 1
Arm/Group | Alisporivir | Boceprevir
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants Who Achieved Sustained Virologic Response (SVR) 24 Weeks After the End of Treatment (SVR24)
Description: SVR24 was defined as hepatitis C virus (HCV) RNA undetectable (by limit of detection) 24 weeks after end of treatment.
Time Frame: 24 weeks post-treatment
Population: as for outcome 1
Arm/Group | Alisporivir | Boceprevir
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Alisporivir: Adverse event (AE) occurred while taking Alisporivir + PEGinf + RBV.
- Boceprevir: AE occurred while taking Boceprevir + PEGinf + RBV.
- PEGinf + RBV: AE occurred while taking only PEGinf + RBV.
- No Intervention: AE was discovered while taking no intervention.
Arm/Group | Alisporivir | Boceprevir | PEGinf + RBV | No Intervention
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 5/5 | 8/8 | 4/8 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisporivir (N=5) | Boceprevir (N=8) | PEGinf + RBV (N=8) | No Intervention (N=6)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alisporivir (N=5) | Boceprevir (N=8) | PEGinf + RBV (N=8) | No Intervention (N=6)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Influenza Like Illness (General disorders) | 1 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Disturbance in Attention (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Haematocrit Decreased (Investigations) | 1 | 1 | 0 | 0
Haemoglobin Decreased (Investigations) | 1 | 1 | 0 | 0
Chest Discomfort (General disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 2 | 0
Libido Decreased (Psychiatric disorders) | 0 | 0 | 2 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Pharyngitis Streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 0 | 1 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 0
Injection Site Erythema (General disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to the early termination of study enrollment and discontinuation of alisporivir treatment, Amendment 1 changed the number of study arms to 2, combining Arms A and B, and none of the planned outcome measures could be evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other